CLINICAL TRIAL: NCT01737853
Title: Comparison of Efficacy and Tolerability Between 2fixed Combinations for Treating Mexican Patients With Primary Open-Angle Glaucoma or Ocular Hypertension: Ganforti vs Krytantek.A Phase IV,Examiner-masked Cross-over Multicenter Clinical Trial
Brief Title: Comparison of Efficacy & Tolerability Between Ganfort vs Krytantek in Mexican Patients With Primary Open-Angle Glaucoma (POAG) or Ocular Hypertension (OHT)
Status: Completed | Type: Observational
Sponsor: Allergan S.A. DE C.V.. (Industry)
Responsible Party: Sponsor
Other Study IDs: ALLE-GANFORT-001-4-2011
Record Dates: First submitted 2012-10-09; First posted 2012-11-30 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-11

CONDITIONS: Glaucoma Primary Open Angle
Keywords: Primary Open-Angle Glaucoma; Ocular Hypertension; Ganfort
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Ganfort

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Ganfort's Group: Ganfort® QD for patients under Krytantek®
  For patients assigned to the Ganfort's group, instructions for applying one drop QD (8:00 PM ± 30 minutes)
  Interventions: Drug: Ganforti
- Krytantek's Group: Krytantek® BID for patients under Ganforti®
  For patients assigned to the Krytantek's group, application schedule will be BID (8:00 AM ± 30 minutes and 8:00 PM ± 30 minutes)
  Interventions: Drug: Krytantek

INTERVENTIONS:
Drug: Ganforti — Enrolled patients will be visiting their clinical site at month 2 and month 3, after starting the study medication; at the end of the third month of treatment, a cross-over maneuver will be indicated; all patients will undergo a follow-up scheme similar to the first period of the study (at month 5 and month 6)
  Other Names: Ganfort
  Groups: Ganfort's Group
Drug: Krytantek — Enrolled patients will be visiting their clinical site at month 2 and month 3, after starting the study medication; at the end of the third month of treatment, a cross-over maneuver will be indicated; all patients will undergo a follow-up scheme similar to the first period of the study (at month 5 and month 6)
  Groups: Krytantek's Group

SUMMARY:
The objective of this phase IV clinical multi-center trial will be to compare the efficacy and safety of Ganforti® versus Krytantek®, using a cross-over design during a six month period (including a one-month wash-in period) in POAG and OH patients.

DETAILED DESCRIPTION:
A prospective examiner-masked, cross-over competitive multicenter clinical trial of 90 consecutive patients derived from three centers in Mexico will be carried out. All eligible eyes should have a diagnosis of either ocular hypertension or mild to moderate POAG with at least 21 mm Hg at baseline (Eligibility Visit), under treatment with either Ganforti® QD or Krytantek® BID. Patients identified to have the selection criteria at the Screening Visit will be scheduled for an Eligibility Visit prior to be prescribed with either of the two study medications (Ganforti® QD for patients under Krytantek®, and Krytantek® BID for patients under Ganforti®). Enrolled patients will be visiting their clinical site at month 2 and month 3, after starting the study medication; at the end of the third month of treatment, a cross-over maneuver will be indicated; all patients will undergo a follow-up scheme similar to the first period of the study (at month 5 and month 6). A battery of tests will be applied in a pre-established regime (table 1). Visual acuity, refraction, biomicroscopy, gonioscopy, dilated fundus examination, Humphrey 24-2 visual field (SITA-Standard), ocular surface fluorescein staining, tear breakup time, OSDI© (Ocular Surface Index) and central ultrasound pachymetry will be administered at baseline and month 6 (at the conclusion of the study). IOP from applanation Goldmann tonometry (8:00 AM ± 1 hour and 10:00 AM ± 1 hour), blood pressure, pulse and a comprehensive ophthalmological examination will be performed at each visit.

Candidate patients will have an initial screening visit where entry criteria must be met (see section 1.7.). Study medication will remain masked to the examiner during the entire trial. For patients assigned to the Ganforti's group, instructions for applying one drop QD (8:00 PM ± 30 minutes); for patients assigned to the Krytantek's group, application schedule will be BID (8:00 AM ± 30 minutes and 8:00 PM ± 30 minutes). Bottles will be given to the patient in a closed labeled box (with the randomization number on it), dispensed by the office assistant, and have to be returned in the same box to the assigned office personnel but never to the principal investigator or sub-investigator, in order to preserve the single-masked nature of the study. New study medication bottles will be dispensed at baseline visit, and monthly after such visit.

Patients will receive verbal instructions, written reminders and periodic phone calls in order to adhere to medication application, as well to scheduled visits (table 1). Outcome variables will also include adverse events (serious, and non-serious, according to the principal investigator's clinical opinion) derived from all examination items. Patient´s and treating ophthalmologist´s subjective satisfaction to the study medication performance will also will be assessed through the closed-end questions (CRF form).

ELIGIBILITY:
Inclusion Criteria:

* Best-corrected visual acuity of at least 20/80 in both eyes
* Age above 17 years
* Use of active contraceptive methods for women in their reproductive phase of life
* Complete demographic and baseline information (Eligibility Visit)
* IOP ≥ 18 mm Hg and ≤ 36 mm Hg
* Significant visual field loss in the previous year
* Uncontrolled systemic disease
* Active ocular disease or intraocular surgery within past three months
* Use of other medications with possible substantial effect on IOP
* Allergy/contraindication to any of the study components
* Severe glaucoma according to Hodapp's criteria
* Incapacity or unwillingness to participate in the study

Exclusion Criteria:

-Any ocular illness other than mild-moderate lens loss of transparency and glaucoma/ocular hypertension

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will enroll 90 patients (45 per treatment group) to yield approximately 80 evaluable patients (40 per treatment group.
  Sample size calculation will take into account the following assumptions:
  * standardized effect size of 0.60
  * 2-sided α value of 0.01 and a β value of 0.10
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2011-02; Primary Completion 2011-02 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
IOP (Intraocular Pressure) | 6 months

SECONDARY OUTCOMES:
Adverse Events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jose A Paczka, MD, Principal Investigator — director of Global Glaucoma Institute; Guadalajara, Jalisco, México.; Karen Ortiz, Study Director — Allergan SA de CV
Locations (4):
- Mexico (4):
  - Global Galucoma Institute, Guadalajara, Jalisco
  - Asociación Para Evitar La Ceguera en México, Mexico City, Mexico City
  - Hospital de Nuestra Señora de la Luz, Mexico City, Mexico City
  - Instituto Oftalmológico Conde de Valencian, Mexico City, Mexico City

REFERENCES:
- [Derived] Garcia-Lopez A, Paczka JA, Jimenez-Roman J, Hartleben C. Efficacy and tolerability of fixed-combination bimatoprost/timolol versus fixed-combination dorzolamide/brimonidine/timolol in patients with primary open-angle glaucoma or ocular hypertension: a multicenter, prospective, crossover study. BMC Ophthalmol. 2014 Dec 19;14:161. doi: 10.1186/1471-2415-14-161. PMID 25527295